CLINICAL TRIAL: NCT00571883
Title: SEND Trial The Role of Selective Neck Dissection Used Electively in Patients With Early Oral Squamous Cell Carcinoma (1-3cm Primary Size) and No Clinical Evidence of Lymph Node Metastases in the Neck
Brief Title: Neck Surgery in Treating Patients With Early-Stage Oral Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Facial Surgery Research Foundation (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000577728; FSRF-SEND-001; EU-20794
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2009-07

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Tongue Neoplasms | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Other: questionnaire administration
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment
Procedure: regional lymph node dissection
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Surgery may be an effective treatment for oral cancer. It is not yet known whether surgery to remove the tumor and lymph nodes in the neck is more effective than surgery to remove the tumor alone in treating patients with early-stage oral cancer.

PURPOSE: This randomized clinical trial is comparing two types of neck surgery to see how well they work in treating patients with early stage oral cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether the use of a selective neck dissection (SEND) used electively on all patients presenting with stage I-II oral cavity squamous cell carcinoma (SCC) improves survival, disease-free survival, and loco-regional disease control rates.
* To determine how SEND and complex reconstruction affect quality of life and mental health.
* To determine whether the use of SEND on all patients presenting with stage I-II oral cavity SCC represents a cost-effective use of resources.

OUTLINE: This is a multicenter study. Patients are stratified by age (< 40 vs 40-64 vs ≥ 65 years of age), tumor stage (T1 vs T2), and surgeon.

* Arm I: Patients undergo resection of the primary tumor with neck dissection.
* Arm II: Patients undergo resection of the primary tumor alone. Patients complete the EORTC QLQ-C30, EORTC QLQ - H&N35, and the Hospital Anxiety and Depression Scale (HADS) before surgery and at 6, 12, and 24 months after surgery. Patients also complete the EQ-5D questionnaire at baseline, 6 months, 12 months, and 24 months. Additionally, a self-completion Health Service Use questionnaire is completed every 2 months, during the first 24 months after treatment, to enable costs to the NHS to be monitored.

After surgery, patients are followed periodically for up to 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with oral squamous cell carcinoma measuring 1 to 3 cm at the primary site
* No clinical or preoperative imaging evidence of nodal involvement in the neck (N0)
* Surgery is the primary mode of treatment

  * Dose not need reconstruction that necessitates opening the neck, as assessed by the surgeon
* No cancer of the lip
* No prior head and neck tumor

PATIENT CHARACTERISTICS:

* No technical, medical, or anaesthetic difficulties that preclude patients being entered into one of the trial arms
* Not considered to be medically, socially, or psychiatrically unfit for surgery as first-line treatment by the multidisciplinary team
* No other synchronous tumor
* No preference for non-surgical treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 652 (Estimated)
Dates: Start 2007-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Disease-free survival
Local and regional recurrence
Completeness of resection at the primary site
Quality-of-life as measured by the EORTC QLQ-30 & H&N module
Psychological well-being as measured by the Hospital Anxiety and Depression Scale (HADS) at 6, 12, and 24 months
Costs to NHS, patients, and carers/families
Incremental cost per life-year saved and/or per quality-adjusted life year (QALY)

CONTACTS AND LOCATIONS:
Overall Officials: Iain Hutchison, Study Chair — The Facial Surgery Research Foundation
Locations (27):
- United Kingdom (27):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Cumberland Infirmary, Carlisle, England
  - Queen Alexandra Hospital, Cosham, England
  - Derbyshire Royal Infirmary, Derby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Leicester Royal Infirmary, Leicester, England
  - Lincoln County Hospital, Lincoln, England
  - Aintree University Hospital, Liverpool, England
  - Facial Surgery Research Foundation, London, England
  - Saint Bartholomew's Hospital, London, England
  - St. George's Hospital, London, England
  - University College of London Hospitals, London, England
  - Luton and Dunstable Hospital, Luton-Bedfordshire, England
  - Wythenshawe Hospital, Manchester, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - Northampton General Hospital, Northampton, England
  - Queen's Medical Centre, Nottingham, England
  - Pennine Acute Hospitals, Oldham, England
  - Queen's Hospital, Romford, England
  - Sunderland Royal Hospital, Sunderland, England
  - Torbay Hospital, Torquay, England
  - New Cross Hospital, Wolverhampton, England
  - Falkirk and District Royal Infirmary, Falkirk, Scotland
  - Southern General Hospital, Glasgow, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - University Hospital of Wales, Cardiff, Wales
  - Barnet General Hospital, Barnet, Hertfordshire

REFERENCES:
- [Derived] Worthington HV, Bulsara VM, Glenny AM, Clarkson JE, Conway DI, Macluskey M. Interventions for the treatment of oral cavity and oropharyngeal cancers: surgical treatment. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD006205. doi: 10.1002/14651858.CD006205.pub5. PMID 37650478
- [Derived] Hutchison IL, Ridout F, Cheung SMY, Shah N, Hardee P, Surwald C, Thiruchelvam J, Cheng L, Mellor TK, Brennan PA, Baldwin AJ, Shaw RJ, Halfpenny W, Danford M, Whitley S, Smith G, Bailey MW, Woodwards B, Patel M, McManners J, Chan CH, Burns A, Praveen P, Camilleri AC, Avery C, Putnam G, Jones K, Webster K, Smith WP, Edge C, McVicar I, Grew N, Hislop S, Kalavrezos N, Martin IC, Hackshaw A. Nationwide randomised trial evaluating elective neck dissection for early stage oral cancer (SEND study) with meta-analysis and concurrent real-world cohort. Br J Cancer. 2019 Nov;121(10):827-836. doi: 10.1038/s41416-019-0587-2. Epub 2019 Oct 15. PMID 31611612